CLINICAL TRIAL: NCT03826901
Title: A Phase 1 Open-label, Multi-centre, Single-arm Trial to Evaluate the Safety and Pharmacokinetics (Including MUsT) of Twice Daily Topical Application of Delgocitinib Cream for 8 Weeks in Adults, Adolescents, and Children With Moderate to Severe Atopic Dermatitis
Brief Title: Delgocitinib Cream for the Treatment of Moderate to Severe Atopic Dermatitis During 8 Weeks in Adults, Adolescents, and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0133-1181
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2021-11

CONDITIONS: Atopic Dermatitis
Keywords: adults, pediatric
MeSH Terms: conditions — Dermatitis, Atopic | interventions — delgocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: adults and adolescents (12 years and above) (Experimental): Delgocitinib cream (dosage: A mg/g).
  Interventions: Drug: delgocitinib
- Part 2: children (2-11 years) (Experimental): Delgocitinib cream (dosage: B mg/g).
  Interventions: Drug: delgocitinib

INTERVENTIONS:
Drug: delgocitinib — Cream for topical application
  Other Names: LEO 124249

SUMMARY:
This is a multi-center, open-label trial to evaluate safety and pharmacokinetics of topical delgocitinib cream applied to pediatric subjects (2-17 years) and adult subjects (18 years and above) with atopic dermatitis.

DETAILED DESCRIPTION:
A phase 1 open-label, multi-centre, single-arm trial to evaluate the safety and pharmacokinetics (including MUsT) of twice daily topical application of delgocitinib cream for 8 weeks in adults, adolescents, and children with moderate to severe atopic dermatitis

ELIGIBILITY:
Key Inclusion criteria (Part 1: adults and adolescents; 12 years and above)

* Diagnosis of atopic dermatitis (AD) as defined by the Hanifin and Rajka (1980) criteria for AD
* Age 12 years and above at baseline
* AD involvement of 25-50% treatable body surface area (BSA) at screening and at baseline
* Moderate to severe AD (Validated Investigator Global Assessment scale for Atopic Dermatitis [vIGA-AD] score of at least 3) at screening and at baseline

Key Inclusion criteria (Part 2: children; 2-11 years)

* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD
* Age 2-11 years at baseline
* History of AD for at least 3 months (children aged 2-5 years), and at least 12 months (children aged 6-11 years)
* AD involvement of ≥35% treatable BSA at screening and at baseline
* Moderate to severe AD (vIGA-AD score of at least 3) at screening and at baseline

Key Exclusion criteria (Part 1 and 2: subjects aged 2 years and above)

* Active dermatologic conditions that may interfere with the diagnosis of AD
* Use of tanning beds or phototherapy within 4 weeks prior to baseline
* Systemic treatment with immunosuppressive/modulating drugs or corticosteroids within 4 weeks prior to baseline or 3 or more bleach baths any week within 4 weeks prior to baseline
* Treatment with topical corticosteroids (TCS), topical calcineurin inhibitors (TCIs), topical phosphodiesterase-4, or oral antibiotics within 1 week prior to baseline
* Clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to baseline
* Any disorder, which is not stable, and in the investigator's opinion could affect the safety of the subject, influence the results of the trial or impede the subject's ability to complete the trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Week 0 to Week 8
  Number of AEs and number of subjects with AEs

SECONDARY OUTCOMES:
PK parameter - Cmax | at Day 8
  Cmax
PK parameter - AUC | at Day 8
  AUC
PK parameter - tmax | at Day 8
  tmax

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (15):
- United States (12):
  - LEO Pharma investigational site, Birmingham, Alabama
  - LEO Pharma investigational site, Phoenix, Arizona
  - LEO Pharma investigational site, Fountain Valley, California
  - LEO Pharma investigational site, Irvine, California
  - LEO Pharma investigational site, Los Angeles, California
  - LEO Pharma investigational site, Centennial, Colorado
  - LEO Pharma investigational site, New Haven, Connecticut
  - LEO Pharma investigational site, Indianapolis, Indiana
  - LEO Pharma investigational site, Ypsilanti, Michigan
  - LEO Pharma investigational site, Tulsa, Oklahoma
  - LEO Pharma investigational site, Medford, Oregon
  - LEO Pharma investigational site, San Antonio, Texas
- Canada (3):
  - LEO Pharma investigational site, Red Deer, Alberta
  - LEO Pharma investigational site, Hamilton, Ontario
  - LEO Pharma investigational site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No